CLINICAL TRIAL: NCT00273624
Title: Olanzapine Augmentation Therapy in Treatment-resistant Depression: a Double-blind Placebo-controlled Trial
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study withdrawn before inclusion of first participant for administrative reasons
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Claus Normann, Prof. Dr., University Hospital Freiburg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Olanzapine Augmentation
Record Dates: First submitted 2006-01-04; First posted 2006-01-09 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Therapy-resistant Depression
Keywords: Therapy-resistant depression; add-on therapy depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- olanzapine (Experimental): 10 mg Olanzapine
  Interventions: Drug: Olanzapine
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Olanzapine — 10 mg Olanzapin concurrent to antidepressive medication
  Other Names: Zyprexa
  Arms: olanzapine
Drug: Placebo — placebo
  Arms: placebo

SUMMARY:
60 patients with major depression will be treated with 10 mg Olanzapine or Placebo for 2 weeks. In case of response (reduction of depressive symptoms)the study will be continued for further 60 days.

DETAILED DESCRIPTION:
The study is using a randomized double-blind, parallel-group, placebo-controlled design. 30 patients per treatment group will be included into the study and randomized to the treatment groups using a computer program. Psychotic features of depression will be excluded by a score of 2 or less in the PANSS subscales P1, P3 and P6. Treatment resistance as defined by history of non-response to two antidepressants from different classes at an acceptable dose and period is confirmed retrospectively. If possible, treatment compliance should be confirmed by plasma level examination. After informed consent, visit 1 is performed on day 0 (inclusion criteria, history, demographics, physical examination, vital signs, HAMD, MADRS, CGI, lab). Study medication is started on day 1, the antidepressive therapy is continued at stable dose until the end of the study. Patients will receive a double-blind therapy of either 10 mg/d olanzapine or placebo. Study visits will be performed on days 4, 7, and 14 (visits 2-4: vital signs, HAMD, MADRS, CGI, lab).

After 14 days, the patients will be classified as responders or non-responders. A responder is defined by a reduction of the initial HAM-D score of more than 50%. Study treatment will be stopped in non-responders and continued in a double-blind manner in responders for further 60 days. Thereafter, the the study medication is stopped and the patients are observed for further 14 days. Study visits will be performed every 14 days. This extension phase was added to examine if a prolonged treatment with olanzapine could ensure a sustained treatment effect. It should be excluded that olanzapine has a short-term tranquillizer-like effect or leads to unfavourable medium- to-long-term depressiogenic effects as observed with other neuroleptics used in depression ( e.g. fluspirilene). Moreover, withdrawal effects should be excluded.

ELIGIBILITY:
Inclusion Criteria:

* major depression without psychotic features
* therapy resistance (2 courses of antidepressants from different classes for more than 3 weeks in adequate dose
* HAM-D score greater/equal than 17
* age 18-65

Exclusion Criteria:

* bipolar disorder
* active alcohol or illicit drug use
* female with ineffective contraception
* severe medical conditions, epilepsy
* psychotic features

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Hamilton-Depression-Scale- HAM-D | 14 days

SECONDARY OUTCOMES:
rate of remission (HAM-D less or equal 7) | 14 days
differences in HAM-D total scores | 14 days
differences in MADRS (Montgomery Asberg Depression Rating Scale)and CGI (Clinical Global Impression)scores | 14 days
predictive value of HAM-D subscales for treatment response use of comedication | 14 days
survival in study | 14 days
differences in rates of adverse events, weight | 14 days
differences in HAM-D scores and survival in extension phase | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Claus Normann, MD, Principal Investigator — Department of Psychiatry, University of Freiburg
Locations (1):
- Dept. of Psychiatry, University of Freiburg, Freiburg im Breisgau, Germany